CLINICAL TRIAL: NCT02952092
Title: A Phase 3, Multi-center, Randomized, 2-arm Parallel, Double-blind, Active-comparator (Darbepoetin Alfa) Conversion Study of Intermittent Oral Dosing of ASP1517 in Hemodialysis Chronic Kidney Disease Patients With Anemia
Brief Title: A Study of Intermittent Oral Dosing of ASP1517 in Hemodialysis Chronic Kidney Disease Patients With Anemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Collaborators: Kyntra Bio (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1517-CL-0307
Record Dates: First submitted 2016-10-31; First posted 2016-11-02 (Estimated); Last update posted 2024-10-30 (Actual); Status verified 2024-10

CONDITIONS: Hemodialysis Chronic Kidney Disease Patients With Anemia
Keywords: ASP1517; Renal anemia; Hemodialysis; Roxadustat
MeSH Terms: interventions — roxadustat; Darbepoetin alfa

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ASP1517 Group (Experimental): Subjects will take the study drug at two- or three-day intervals.
  Interventions: Drug: roxadustat
- Darbepoetin alfa Group (Experimental): Subjects will take the study drug once a week.
  Interventions: Drug: Darbepoetin alfa

INTERVENTIONS:
Drug: roxadustat — Oral
  Other Names: ASP1517
  Arms: ASP1517 Group
Drug: Darbepoetin alfa — Intravenous
  Arms: Darbepoetin alfa Group

SUMMARY:
The objective of this study is to evaluate the safety and efficacy of ASP1517 compared to darbepoetin alfa in hemodialysis chronic kidney disease patients with anemia.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with renal anemia who have been receiving recombinant human erythropoietin (rHuEPO, two times weekly or three times weekly) or darbepoetin alfa (intravenous treatment) within the doses approved in Japan for more than 8 weeks before the screening assessment
* Mean of the subject's two most recent Hb values before dialysis after the longest dialysis interval during the Screening Period must be ≥10.0 g/dL and ≤12.0 g/dL
* Either transferrin saturation (TSAT) ≥ 20% or serum ferritin ≥ 100 ng/mL during the screening period
* Female subject must either:

Be of non-childbearing potential:

* post-menopausal (defined as at least 1 year without any menses) prior to Screening, or
* documented surgically sterile Or, if of childbearing potential,
* Agree not to try to become pregnant during the study and for 28 days after the final study drug administration
* And have a negative pregnancy test at Screening
* And, if heterosexually active, agree to consistently use two forms of highly effective form of birth control (at least one of which must be a barrier method) starting at Screening and throughout the study period and continued for 28 days after the final study drug administration.

  * Female subject must agree not to breastfeed starting at Screening and throughout the study period, and continued for 28 days after the final study drug administration.
  * Female subject must not donate ova starting at Screening and throughout the study period, and continued for 28 days after the final study drug administration.
  * Male subject and their female spouse/partners who are of childbearing potential must be using two forms of highly effective form of birth control (at least one of which must be a barrier method) starting at Screening and continue throughout the study period, and for 12 weeks after the final study drug administration
  * Male subject must not donate sperm starting at Screening and throughout the study period and, for 12 weeks after the final study drug administration

Exclusion Criteria:

* Concurrent retinal neovascular lesion untreated and macular edema untreated
* Concurrent autoimmune disease with inflammation that could impact erythropoiesis
* History of gastric/intestinal resection considered influential on the absorption of drugs in the gastrointestinal tract (excluding resection of gastric or colon polyps) or concurrent gastroparesis
* Uncontrolled hypertension
* Concurrent congestive heart failure (NYHA Class III or higher)
* History of hospitalization for treatment of stroke, myocardial infarction, or pulmonary embolism within 12 weeks before the screening assessment
* Positive for hepatitis B surface antigen (HBsAg) or anti-hepatitis C virus (HCV) antibody at the screening assessment, or positive for human immunodeficiency virus (HIV) in a past test
* Concurrent other form of anemia than renal anemia
* History of pure red cell aplasia
* Having received treatment with protein anabolic hormone, testosterone enanthate, or mepitiostane within 6 weeks before the screening assessment
* Aspartate Aminotransferase (AST), Alanine Aminotransferase (ALT), or total bilirubin that is greater than the criteria, or previous or concurrent another serious liver disease at screening assessment
* Previous or current malignant tumor (no recurrence for at least 5 years is eligible.)
* Having undergone blood transfusion and/or a surgical procedure considered to promote anemia (excluding shunt reconstruction surgery for access to the blood) and/or ophthalmological surgery within 4 weeks before the screening assessment
* Having undergone a kidney transplantation
* Having a previous history of treatment with ASP1517
* History of serious drug allergy including anaphylactic shock
* Participation in another clinical study or post-marketing clinical study (including that of a medical device) within 12 weeks before informed consent acquisition

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 303 (Actual)
Dates: Start 2016-11-30 (Actual); Primary Completion 2018-03-13 (Actual); Study Completion 2018-03-15 (Actual)

PRIMARY OUTCOMES:
Change from baseline in the average hemoglobin (Hb) | Baseline and Weeks 18 to 24

SECONDARY OUTCOMES:
Average Hb from Week 18 to Week 24 | Week 18 to 24
Proportion of participants with the target Hb level from Week 18 to Week 24 | Week 18 to 24
Proportion of participants with the target Hb level at each week | Up to Week 24
Change from week 0 in Hb levels to each week | Up to Week 24
Proportion of measurement points with the target Hb level from Week 18 to Week 24 | Week 18 to 24
Rate of rise in Hb levels (g/dL/week) from week 0 to at the earliest date of week 4, time of discontinuation, or time of dose adjustment | Up to Week 4
Average hematocrit level | Up to Week 24
Average reticulocyte level | Up to Week 24
Average iron (Fe) level | Up to Week 24
Average ferritin level | Up to Week 24
Average transferrin level | Up to Week 24
Average total iron binding capacity level | Up to Week 24
Average soluble transferrin receptor level | Up to Week 24
Average transferrin saturation level | Up to Week 24
Average reticulocyte hemoglobin content level | Up to Week 24
Quality of life assessed by SF-36 | Up to Week 24
  SF-36: Medical Outcomes Study 36-Item Short-Form Health Survey
Quality of life assessed by EQ-5D-5L | Up to Week 24
  EQ-5D-5L: EuroQol 5 Dimension 5-Levels
Quality of life assessed by FACT-An | Up to Week 24
  FACT-An: Functional Assessment of Cancer Therapy-Anemia
Number of hospitalizations | Up to Week 24
Duration of hospitalizations | Up to Week 24
Plasma concentration of unchanged ASP1517 | Up to Week 24
Safety assessed by incidence of adverse events | Up to Week 24
Number of participants with abnormal Laboratory values and/or adverse events related to treatment | Up to Week 24
Number of participants with abnormal Vital signs and/or adverse events related to treatment | Up to Week 24
Number of participants with abnormal 12-lead electrocardiogram (ECG) values | Up to Week 24
  Any clinically significant adverse changes on the ECG will be reported as adverse events.
Safety assessed by ophthalmological examination: fundoscopy | Up to Week 24
Safety assessed by ophthalmological examination: Optical coherence tomography | Up to Week 24
Safety assessed by ophthalmological examination: visual acuity | Up to Week 24

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Inc
Locations (57):
- Japan (57):
  - Site JP00008, Aichi
  - Site JP00018, Aichi
  - Site JP00020, Aichi
  - Site JP00032, Aichi
  - Site JP00033, Aichi
  - Site JP00040, Aichi
  - Site JP00004, Ehime
  - Site JP00055, Ehime
  - Site JP00009, Fukui
  - Site JP00059, Fukui
  - Site JP00014, Fukuoka
  - Site JP00049, Fukuoka
  - Site JP00010, Fukushima
  - Site JP00056, Fukushima
  - Site JP00057, Fukushima
  - Site JP00030, Gifu
  - Site JP00050, Gifu
  - Site JP00011, Gunma
  - Site JP00026, Gunma
  - Site JP00037, Gunma
  - Site JP00003, Hokkaido
  - Site JP00031, Hokkaido
  - Site JP00038, Hokkaido
  - Site JP00048, Hokkaido
  - Site JP00017, Ibaraki
  - Site JP00041, Ibaraki
  - Site JP00042, Ibaraki
  - Site JP00045, Ibaraki
  - Site JP00046, Ibaraki
  - Site JP00047, Ibaraki
  - Site JP00054, Ibaraki
  - Site JP00058, Ibaraki
  - Site JP00043, Kagoshima
  - Site JP00005, Kanagawa
  - Site JP00028, Kumamoto
  - Site JP00029, Kumamoto
  - Site JP00006, Kyoto
  - Site JP00002, Nagano
  - Site JP00012, Nagano
  - Site JP00027, Nagano
  - Site JP00051, Nagano
  - Site JP00013, Nagasaki
  - Site JP00001, Niigata
  - Site JP00034, Niigata
  - Site JP00036, Okayama
  - Site JP00007, Osaka
  - Site JP00015, Osaka
  - Site JP00016, Saitama
  - Site JP00035, Saitama
  - Site JP00044, Tokushima
  - Site JP00052, Tokyo
  - Site JP00053, Tokyo
  - Site JP00021, Toyama
  - Site JP00022, Toyama
  - Site JP00039, Toyama
  - Site JP00024, Yamagata
  - Site JP00025, Yamaguchi

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.

REFERENCES:
- [Derived] Hamano T, Yamaguchi Y, Goto K, Mizokawa S, Ito Y, Dellanna F, Barratt J, Akizawa T. Risk Factors for Thromboembolic Events in Patients With Dialysis-Dependent CKD: Pooled Analysis of Phase 3 Roxadustat Trials in Japan. Adv Ther. 2024 Apr;41(4):1526-1552. doi: 10.1007/s12325-023-02727-3. Epub 2024 Feb 16. PMID 38363463
- [Derived] Natale P, Palmer SC, Jaure A, Hodson EM, Ruospo M, Cooper TE, Hahn D, Saglimbene VM, Craig JC, Strippoli GF. Hypoxia-inducible factor stabilisers for the anaemia of chronic kidney disease. Cochrane Database Syst Rev. 2022 Aug 25;8(8):CD013751. doi: 10.1002/14651858.CD013751.pub2. PMID 36005278
- [Derived] Akizawa T, Iwasaki M, Yamaguchi Y, Majikawa Y, Reusch M. Phase 3, Randomized, Double-Blind, Active-Comparator (Darbepoetin Alfa) Study of Oral Roxadustat in CKD Patients with Anemia on Hemodialysis in Japan. J Am Soc Nephrol. 2020 Jul;31(7):1628-1639. doi: 10.1681/ASN.2019060623. Epub 2020 Jun 3. PMID 32493693
- See also: Link to results on Astellas Clinical Study Results website — https://astellasclinicalstudyresults.com/study.aspx?ID=356